CLINICAL TRIAL: NCT02270632
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Study to Evaluate Safety and Clinical Efficacy of Two Different Doses of F8IL10 (Dekavil) Administered Subcutaneously to Patients With Active Rheumatoid Arthritis Receiving Methotrexate.
Brief Title: A Randomized, Placebo-controlled Phase II Clinical Trial to Evaluate the Safety and Efficacy of F8IL10 (Dekavil) in Patients With Active RA Receiving MTX
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Approvals of new agents for the same indication have significantly slowed down the recruitment in this trial making the prosecution of the present investigation extremely difficult.
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PH-F8IL10-03/13
Record Dates: First submitted 2014-10-16; First posted 2014-10-21 (Estimated); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Placebo Comparator): Placebo
  Interventions: Drug: MTX; Drug: Placebo
- Arm 2 (Experimental): F8IL10, 30 μg/kg
  Interventions: Drug: F8IL10; Drug: MTX
- Arm 3 (Experimental): F8IL10, 160 μg/kg
  Interventions: Drug: F8IL10; Drug: MTX

INTERVENTIONS:
Drug: F8IL10 — F8IL10 will be administered once a week for 8 weeks (or until withdrawn from the study).
  Other Names: Dekavil
  Arms: Arm 2; Arm 3
Drug: MTX — All patients enrolled in the study will receive as concomitant therapy MTX at stable dose (10-25 mg/week), and the corresponding fixed dose of folic acid.
  Other Names: Methotrexate
Drug: Placebo — Placebo will be administered once a week for 8 weeks (or until withdrawn from the study).
  Arms: Arm 1

SUMMARY:
A multicenter, randomized, parallel assignment, double blind, placebo-controlled, safety/efficacy phase II study of two different dosages of subcutaneous F8IL10 in patients with active rheumatoid arthritis receiving MTX.

DETAILED DESCRIPTION:
The study is designed to formally demonstrate the superiority of F8IL10 vs placebo and to further evaluate safety and efficacy of two different dosages of F8IL10 when administered to patients receiving MTX.

Patients will be enrolled and double-blind, parallel assigned (via automated randomization system) in a 1:1:1 fashion to one of three different arms:

* Arm 1: placebo + MTX
* Arm 2: F8IL10 30 µg/kg + MTX
* Arm 3: F8IL10 160 µg/kg + MTX

F8IL10 or placebo will be subcutaneously injected once a week for 8 weeks. Treatment will terminate at the earliest of the following: completion of the 8 weeks of therapy, withdrawal of informed consent, unacceptable toxicity/intolerability of the study drug or need to increase MTX, oral corticosteroids or NSAIDs dosages above baseline levels or need to introduce a new DMARD or biologic therapy to control rheumatoid arthritis activity. The study will be conducted in a double blind fashion.

ELIGIBILITY:
Inclusion Criteria

At the time of enrolment, patients must fulfil all of the following criteria:

1. Patients aged ≥18 and < 75 years.
2. Diagnosis of RA according to ACR/EULAR classification criteria (2010) with a disease duration exceeding 6 months.
3. Active RA (DAS28 ≥ 3.2) for ≥ 3 months at time of signing informed consent despite MTX therapy (stable regimen of methotrexate 10-25 mg/week orally, subcutaneous or intramuscular injections: stable dosage from ≥ 8 weeks before screening).
4. ≥ 6 tender joints out of 68, ≥ 6 swollen joints out of 66 and serum CRP > 0.5 mg/dl at screening.
5. History of inadequate clinical response to at least one anti-TNF drug (applied for at least 3 months).
6. Stable regimens of NSAIDs and/or oral corticosteroid (≤ 10 mg/day; prednisone equivalent) for a period ≥ 2 weeks prior to screening.
7. All acute toxic effects of any prior therapy must have returned to classification "mild" according to CTCAE v.4.03 (published on June 14, 2010).
8. Sufficient hematologic, liver and renal function:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelets ≥100 x109/L, haemoglobin (Hb) ≥ 10.0 g/dL.
   * Alkaline phosphatase (AP), alanine aminotransferase (ALT) and or aspartate aminotransferase (AST) ≤ 3 x upper limit of normal range (ULN), and total bilirubin ≤ 2.0 mg/dl (34.2 µmol/L).
   * Creatinine ≤ 1.5 ULN or 24 h creatinine clearance ≥ 50 mL/min.
9. Documented negative test for HIV, HBV and HCV. For patients with serology documenting previous exposure to HBV (i.e., anti-HBs Ab with no history of vaccination and/or anti-HBc Ab), negative serum HBV DNA is required.
10. All female subjects must have negative pregnancy test results at the screening. Women of childbearing potential must be using simultaneously double-barrier or two acceptable methods of contraception (i.e. intra-uterine device plus condom, spermicidal gel plus condom, diaphragm plus condom, etc.) from the screening to three months following the last study drug administration. Pregnancy test will be repeated at the end of treatment visit.
11. Male patients must agree to use simultaneously two acceptable methods of contraception (i.e. spermicidal gel plus condom) from the screening to three months following the last study drug administration.
12. Signed and dated Ethics Committee-approved informed consent form indicating that the patient has been informed of all pertinent aspects of the study.
13. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.
14. Chest X rays performed (for other reasons than the present clinical trial) within a period of 3 months prior to the screening visit. However, in the case the patient performs the Quantiferon TB test during the screening visit, this period can be extended to 6 months.

Exclusion Criteria

Patients must not be enrolled into the study if, at the time of enrolment, they have any of the following:

1. Presence of active infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or would interfere with the study objectives or conduct.
2. Pregnancy, lactation or unwillingness to use adequate contraceptive methods.
3. Diagnosis of any other inflammatory arthritis or active autoimmune diseases other than RA.
4. Last treatment with monoclonal antibodies (i.e., adalimumab, infliximab, golimumab, tocilizumab, certolizumab pegol) less than 8 weeks prior to first administration of study drugs. Last treatment with rituximab less than 16 weeks prior to first administration of study drugs. Last treatment with fusion proteins (i.e., abatacept, etanercept) less than 4 weeks prior to first administration of study drugs.
5. Treatment with any immunosuppressant drug other than MTX and corticosteroids.
6. Active or latent tuberculosis (TB).
7. HIV infection.
8. Acute or chronic HBV or HCV infection, as assessed by serology or serum HBV DNA.
9. History or currently active primary or secondary immunodeficiency.
10. Concurrent malignancy or history of malignancy from which the patient has been disease-free for less than 5 years.
11. History within the last year of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
12. Treatment with warfarin or other coumarin derivatives.
13. Heart insufficiency (> Grade II, NYHA criteria).
14. Irreversible cardiac arrhythmias requiring permanent medication.
15. Clinically significant (to clinical investigator's discretion) abnormalities in baseline ECG analysis.
16. Uncontrolled hypertension.
17. Ischemic peripheral vascular disease (Grade IIb-IV).
18. Severe diabetic retinopathy.
19. Major trauma including surgery within 4 weeks prior to administration of study treatment.
20. Known history of allergy or other intolerance to IL10, methotrexate, folic acid or other drugs based on human proteins/peptides/antibodies.
21. Treatment with any investigational agent within the 6 weeks before study treatment.
22. Immunization with a live/attenuated vaccine within 4 weeks prior to baseline or plan to receive vaccines during the study.
23. Treatment with growth factors or immunomodulatory agents, including Anakinra, within 7 days of the administration of study drugs.
24. Chronic pain disorders (not RA-related) that might interfere with pain evaluation.
25. Patients requiring stable doses of corticosteroids > 10 mg/day (prednisone equivalent). Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions is not considered an exclusion criterion.
26. Concurrent intra-articular corticosteroids treatment or patient who have received it within 2 weeks prior to randomization.
27. History of alcohol, drug or chemical substance abuse within the 6 months prior to screening.
28. Any condition that in the opinion of the investigator could hamper compliance with the study protocol.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in DAS28-CRPscore | At week 9
  Mean change from baseline in DAS28-CRP between F8IL10 and placebo arms.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | Up to 8 months from randomization
  Safety and tolerability of subcutaneous F8IL10 when administered in combination with MTX.
Response rate according to ACR and EULAR criteria | 1) week 9; 2) from week 12 up to week 32, every 4 weeks
  Proportion of patients achieving an ACR clinical response (ACR20, 50 and 70) and time to onset of these criteria.
Clinical Remission and low-disease activity (DAS28-CRP) | 1) week 9; 2) from week 12 up to week 32, every 4 weeks
  Proportion of patients achieving clinical remission and clinical low- disease activity according to DAS 28-CRP (DAS28 < 2.6 and 2.6≤ DAS28 <3.2, respectively) and time to onset of these criteria.
Clinical Remission and low-disease activity (SDAI score) | 1) week 9; 2) from week 12 up to week 32, every 4 weeks
  Proportion of patients achieving clinical remission and clinical low-disease activity according to SDAI score (SDAI ≤ 3.3 and SDAI ≤ 11.0) and time to onset of these criteria
Absolute count and change from baseline in tender and swollen joint counts | 1) from week 1 up to week 9; 2) from week 12 up to week 32, every 4 weeks
  The tender joint count represents the number of joints in which pain is reported at rest with pressure or on movement.
  The swollen joint count represents the number of joints in which there is synovial fluid and/or soft tissue swelling.
Absolute score and change from baseline in physician's and patient's global assessments of disease activity (100 mm VAS) | 1) from week 1 up to week 9; 2) from week 12 up to week 32, every 4 weeks
  Patient's and Physician's global assessment of disease activity.
Absolute score and change from baseline in patient assessment of the pain intensity at each visit (100 mm VAS) | 1) from week 1 up to week 9; 2) from week 12 up to week 32, every 4 weeks
  Patient's assessment of pain.
Proportion of patients that experienced significant change from baseline in functional status (HAQ-DI) | 1) week 9; 2) from week 12 up to week 32, every 4 weeks
Proportion of patients that experienced significant change from baseline in functional status (SF-36) | 1) week 9; 2) from week 12 up to week 32, every 4 weeks
HAQ score and change from baseline in HAQ score | 1) week 1; 2) week 9; 3) from week 12 up to week 32, every 4 weeks
Inflammatory parameters CRP or ESR and change from baseline | 1) from week 1 up to week 9; 2) from week 12 up to week 32, every 4 weeks
  Laboratory assessments (CRP, ESR)
Human anti-fusion protein antibodies (HAFA) levels | 1) day 14 - 0 (screening); 2) at week 1; 3) at week 5; 4) at week 9 (EoT); 5) from week 12 up to week 32, every 4 weeks
  Investigate the potential induction of human anti-fusion protein antibodies (HAFA) through standard laboratory analysis.
Percentage of Participants With Worst On-Study Hematological and Chemistry Abnormalities | 1) from week 1 up to week 9; 2) from week 12 up to week 32, every 4 weeks
Clinically Meaningful Changes in Vital Signs and Physical Examinations | 1) from week 1 up to week 9; 2) from week 12 up to week 32, every 4 weeks
Changes in absolute counts and relative percentages of main biomarker/cytokines | 1) day 14 - 0 (screening); 2) at week 1; 3) at week 5; 4) at week 9 (EoT); 5) from week 12 up to week 32, every 4 weeks
  Biomarkers :IgA, IgE, Soluble IL-2 receptor, Soluble IL-1 receptor antagonist, MMP3); cytokines: IL-1α, IL-1β, TNFα, IL2, IL6, IL17, IL18, IL22, VEGF

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (3):
  - Universitatsklinikum Essen, Essen
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Schön Klinik Hamburg Eilbek, Hamburg
- Italy (3):
  - Ospedale Luigi Sacco, Milano, Milan
  - Azienda Ospedaliera Universitaria Senese, Siena
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Switzerland (2):
  - HFR Fribourg - Hôpital Cantonal, Fribourg
  - Centre Hospitalier Universitaire Vaudois, Lausanne